CLINICAL TRIAL: NCT04704635
Title: The Relationship Between Trajectories of Post-stroke Disability and Self-rated Health
Brief Title: Trajectories of Post-stroke Multidimensional Health
Acronym: NeuroAdapt
Status: Completed | Type: Observational
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Principal Investigator, Susanne Wurm, Principal Investigator, Head of Prevention Research and Social Medicine, University Medicine Greifswald
Other Study IDs: NeuroAdapt
Record Dates: First submitted 2021-01-08; First posted 2021-01-11 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Stroke, Ischemic; Transient Ischemic Attack; Adaptation, Psychological; Mental Health Impairment; Adjustment; Self-Rated Health; Aging; Sense of Coherence
Keywords: Old Age; Mental Health; Psychological Health; Self-Rated Health; Quality of Life; Views on Aging; Resilience; Salutogenesis
MeSH Terms: conditions — Ischemic Stroke; Ischemic Attack, Transient; Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ischemic stroke/TIA: Patients with ischemic stroke or transient ischemic attack

SUMMARY:
Stroke is thought to cause disability immediately after stroke followed by a 3-to-6-month recovery period, after which disability levels are supposed to stabilize unless recurrent events occur. However, studies showed that post-stroke recovery is heterogeneous. While some stroke survivors quickly recover, others may show an accelerated accumulation of disability over time. The current prospective observational study will investigate trajectories of multidimensional functioning and self-rated health in the year after stroke. Particularly, the study aims to explore the relationship between trajectories of disability and self-rated health. Moreover, the study will focus on potential predictors of changes in disability and self-rated health, i.e., views on aging and psychological resilience. Patients will be recruited during their stay at the stroke unit and participate in a face-to-face interview and four follow-up telephone interviews in the post-stroke year.

DETAILED DESCRIPTION:
Ischemic strokes have shown to have long-term impact on functional health apart from their acute effects on neurological functioning. Stroke survivors may experience long-term physical disability, psychopathological symptoms and cognitive decline. Even though these potential consequences are well studied, knowledge on post-stroke trajectories of multidimensional functional health according to the Word Health Organization's (WHO) International Classification of Functioning, Disability and Health (ICF) and their predictors is rare. Particularly, there is a lack of studies investigating the trajectories of self-rated health and different indicators of functional health in the year post-stroke. Therefore, the current study aims to explore trajectories of disability and self-rated health in the year post-stroke, and is the first to analyze the relationship between these trajectories. Thereby, the study addresses the research question whether changes in disability can be predicted by prior self-rated health or changes of self-rated health, and vice versa. Moreover, the study examines the correspondence between changes of disability and self-rated health in the year post-stroke. Additionally, views on aging and psychological resilience, which are relevant to coping processes, are studied as predictors of changes in disability and self-rated health. Patients recruited during their stay at the stroke unit will participate in one face-to-face interview in hospital and four telephone follow-up interviews at 6 weeks, 3 months, 6 months and 12 months post-stroke. Moreover, physical functioning will be externally assessed during their hospital stay. To increase the knowledge on post-stroke trajectories of multidimensional health is of major importance to identify patients at risk for accelerated accumulation of disability. Findings from the current study may contribute to the improvement of post-stroke rehabilitation and secondary prevention.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50 years
* Acute ischemic stroke/high-risk transient ischemic attack (TIA; ABCD2 score ≥ 3)
* Language: Fluent in German
* Written informed consent of patient or caregiver

Exclusion Criteria:

* Low-risk TIA (ABCD2 score ≤ 2)
* Severe cognitive impairment (i.e., incomplete orientation)
* Severe communication disorder
* Index event > 5 days prior to enrolment
* Life expectancy < 1 year

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with acute ischemic stroke/transient ischemic attack (TIA) are enrolled during their acute treatment (1-5 days post-acute ischemic stroke/TIA). Patients with an ABCD2 score ≤ 2 are excluded to reduce the chance of inclusion of patients with TIA mimic. The number of TIA patients is limited to 20% of the sample to avoid a bias towards TIA and to represent common incidents of acute ischemic stroke.
Sampling Method: Non-Probability Sample
Enrollment: 330 (Actual)
Dates: Start 2021-05-12 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2023-09-18 (Actual)

PRIMARY OUTCOMES:
Change of Modified Rankin Scale (self-reported) | 1-5 days post-stroke, 6 weeks post-stroke, 3 months post-stroke, 6 months post-stroke, 12 months post-stroke
  Degree of disability and dependency
Change of self-rated health | 1-5 days post-stroke, 6 weeks post-stroke, 3 months post-stroke, 6 months post-stroke, 12 months post-stroke
  1-Item assessment of self-rated health

SECONDARY OUTCOMES:
Change of Barthel Index (self-reported) | 1-5 days post-stroke, 6 weeks post-stroke, 3 months post-stroke, 6 months post-stroke, 12 months post-stroke
  Measure of performance in activities of daily living
Change of Impact of Stroke Scale 16 | 1-5 days post-stroke, 6 weeks post-stroke, 3 months post-stroke, 6 months post-stroke, 12 months post-stroke
  Assessment of the impact of stroke on four domains (i.e., strength, hand function, mobility, and activities of daily living)
Change of European Health Interview Survey Physical Activity Questionnaire | 1-5 days post-stroke, 6 weeks post-stroke, 3 months post-stroke, 6 months post-stroke, 12 months post-stroke
  Assessment of physical activity
Change of European Quality of Life 5 Dimensions 5 Level Version (EQ-5D-5L) | 1-5 days post-stroke, 6 weeks post-stroke, 3 months post-stroke, 6 months post-stroke, 12 months post-stroke
  Assessment of quality of life
Change of IMET (Index for the Assessment of Participation Restrictions) | 1-5 days post-stroke, 6 weeks post-stroke, 3 months post-stroke, 6 months post-stroke, 12 months post-stroke
  Assessment of restrictions of participation (according to the WHO concept)
Change of Fatigue Severity Scale | 1-5 days post-stroke, 6 weeks post-stroke, 3 months post-stroke, 6 months post-stroke, 12 months post-stroke
  Assessment of fatigue
Change of Patient Health Questionnaire-8 | 1-5 days post-stroke, 6 weeks post-stroke, 3 months post-stroke, 6 months post-stroke, 12 months post-stroke
  Assessment of depressive symptoms
Change of Pittsburgh Sleep Quality Index (assessment in case of sufficient capacities) | 1-5 days post-stroke, 6 weeks post-stroke, 3 months post-stroke, 6 months post-stroke, 12 months post-stroke
  Assessment of sleep quality (3 items)
Change of Post-Traumatic Stress Syndrome 14 (assessment in case of sufficient capacities) | 6 weeks post-stroke, 3 months post-stroke, 6 months post-stroke, 12 months post-stroke
  Assessment of posttraumatic stress symptoms
Change of Questions on Falling | 1-5 days post-stroke, 6 weeks post-stroke, 3 months post-stroke, 6 months post-stroke, 12 months post-stroke
  5 items on falls and fear of falling

OTHER OUTCOMES:
Change of SHARE FI | 1-5 days post-stroke, 6 weeks post-stroke (no GSA), 3 months post-stroke (no GSA), 6 months post-stroke (no GSA), 12 months post-stroke (no GSA)
  Assessment of Frailty including grip strength assessment (GSA)
Change of Brief-Illness Perception Questionnaire | 1-5 days post-stroke, 6 weeks post-stroke, 3 months post-stroke, 6 months post-stroke, 12 months post-stroke
  Assessment of illness perceptions
Change of De Jong Gierveld Loneliness Scale (assessment in case of sufficient capacities) | 1-5 days post-stroke, 6 weeks post-stroke, 3 months post-stroke, 6 months post-stroke, 12 months post-stroke
  Assessment of feelings of loneliness
Change of subjective age | 1-5 days post-stroke, 6 weeks post-stroke, 3 months post-stroke, 6 months post-stroke, 12 months post-stroke
  Assessment of subjective age
Change of AgeCog Scales | 1-5 days post-stroke, 6 weeks post-stroke, 3 months post-stroke, 6 months post-stroke, 12 months post-stroke
  Assessment of self-perception of aging
Change of SOK (Selection, Optimization, Compensation) | 1-5 days post-stroke, 6 weeks post-stroke, 3 months post-stroke, 6 months post-stroke, 12 months post-stroke
  Assessment of healthy lifestyle
Change of social support (assessment in case of sufficient capacities) | 1-5 days post-stroke, 6 weeks post-stroke, 3 months post-stroke, 6 months post-stroke, 12 months post-stroke
  Assessment of social support (GEDA/EHIS)
Change of Resilience Scale 13 (assessment in case of sufficient capacities) | 1-5 days post-stroke, 12 months post-stroke
  Assessment of trait-resilience
Change of Brief Assessment of Sense of Coherence | 1-5 days post-stroke, 6 weeks post-stroke, 3 months post-stroke, 6 months post-stroke, 12 months post-stroke
  Assessment of sense of coherence
Change of Generalized Self-Efficacy Scale | 1-5 days post-stroke, 12 months post-stroke
  Assessment of self-efficacy (4 items)
Change of Posttraumatic Growth Inventory (assessment in case of sufficient capacities) | 6 weeks post-stroke, 3 months post-stroke, 6 months post-stroke, 12 months post-stroke
  Assessment of posttraumatic growth (10 items)

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Flöel, PhD, Principal Investigator — University Medicine Greifswald; Robert Fleischmann, PhD, Principal Investigator — University Medicine Greifswald; Bettina von Sarnowski, PhD, Principal Investigator — University Medicine Greifswald
Locations (1):
- University Medicine Greifswald, Greifswald, Germany

REFERENCES:
- [Derived] Schafer SK, Fleischmann R, von Sarnowski B, Blasing D, Floel A, Wurm S. Relationship between trajectories of post-stroke disability and self-rated health (NeuroAdapt): protocol for a prospective observational study. BMJ Open. 2021 Jun 29;11(6):e049944. doi: 10.1136/bmjopen-2021-049944. PMID 34187831